CLINICAL TRIAL: NCT02271490
Title: Improvement of the Post ICSI Pregnancy Outcome by Induction of the Acrosome Reaction Prior to ICSI
Brief Title: Acrosome Reaction Induction Prior to ICSI
Acronym: RA-ICSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-A01376-35
Record Dates: First submitted 2014-10-07; First posted 2014-10-22 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Assisted Reproductive Technique; ICSI; Acrosome Reaction; Pregnancy Outcome
Keywords: Assisted Reproductive Technique; ICSI; Acrosome Reaction; Pregnancy outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- micoinjection according to classical protocole (Active Comparator): incubation of sperm in incubation medium
  Interventions: Other: capacitation in incubation medium prior to ICSI
- incubation in follicular fluid (Experimental): incubation of sperm in follicular fluid prior to microinjection
  Interventions: Other: Acrosome Reaction induction

INTERVENTIONS:
Other: Acrosome Reaction induction
  Arms: incubation in follicular fluid
Other: capacitation in incubation medium prior to ICSI
  Arms: micoinjection according to classical protocole

SUMMARY:
Introduction To get through the egg vestment and fertilize the oocyte, the spermatozoon uses its acrosomal enzymes. When Intracytoplasmic sperm microinjection (ICSI) is performed, the acrosomal enzymes are introduced with the spermatozoa inside the ooplasme.

The fate of these enzymes, that normally never enter the oocyte, is not known. But they impair the embryo development.

Indeed, although the ICSI outcome is satisfactory in humans, a series of studies in many species (mouse, hamster, cattle, and horse) demonstrate the deleterious effects of the introduction of acrosomal material in the oocyte cytoplasm, on embryo and fetal development. These studies have also shown two things:

* The bigger the acrosome, the more deleterious are the effects of their introduction into the egg.
* And that the induction of the acrosome reaction (AR) prior to ICSI significantly improves embryonic development and the number of babies born after embryo transfer as it is the case in the mouse. The microinjection of acrosome reacted sperm increases from 40 to 70 % the percentage of pups born per embryo transferred.

Hypothesis :

It is possible to improve ICSI outcome, in terms of babies born in human, by induction of the AR prior to microinjection.

After studying several techniques, we choose a physiologic technique for acrosome induction.

The induction of acrosome reaction prior to ICSI should improve in utero fetal development and decrease the rate of miscarriage and pregnancy arrest.

DETAILED DESCRIPTION:
1. Introduction Intracytoplasmic sperm microinjection (ICSI) produces 70% of fertilized oocytes and zygotes which mostly develop normally. To perform ICSI, a spermatozoon is taken from a sperm suspension after gradient migration. It is then immobilized by breaking its flagellum using a micropipette, and introduced into the oocyte cytoplasm.

   The rate of spontaneous acrosome reaction in humans is less than 20 %. Two studies on the percentage of acrosome reacted and immobilized sperm showed that 95% of them have a destabilization of the membrane but only 17.8% of them had made a full RA. In other words, when we microinjected 10 spermatozoa, only 2 of them are completely rid of their acrosome material. All others are introduced into the oocyte with acrosomal material. But this material does not normally enter the oocyte since the acrosome reaction is a prerequisite to the passage of the zona pellucida that surrounds the egg .

   The importance of using an acrosome-reacted spermatozoon for the success of ICSI has been previously highlighted in several animal species. It has been demonstrated that the induction of the acrosome reaction in mice lead to higher fertilization rates (from 30% to about 60 % ) . It is similar, in the rabbit and horses . Kimura et al. also reported that mouse oocytes injected with acrosome-intact rabbit and hamster sperm exhibited a nuclear activation and cessation of embryonic development without reaching the two-cell stage. This "cytotoxicity" of the same sperm disappears when they are released from their acrosomes before injection. In another study, the detrimental effect on oocyte survival of the presence of the acrosome during the injection of sperm heads was demonstrated in the golden hamster. All oocytes microinjected with acrosome-intact sperm were dead, while only those injected with acrosome reacted sperm have not only survived, but have also developed to the stage of two pronucleus in 79 % of cases and helped to get live births ( 19%).

   The team of Yanagimachi reported a study on the potentially dangerous effect of the incorporation of the sperm acrosome of different species within mouse oocytes. According to these authors, harmful components would probably be the enzymes such as trypsin-like acrosine and hyaluronidase, since their injection mimicked the effects of ICSI with acrosome-intact sperm. In the same study, it was confirmed that the toxic effects were correlated with the size of the acrosome and therefore the contents of protease enzymes.

   The toxic effects of the acrosome and its contents have been described explicitly by Morozumi and Yanagimachi. It induces deformation of the oocyte with an irregular appearance, edema or cytolysis with a pseudo-vacuolated cytoplasm appearance. Furthermore, it has been established that the damage caused by exogenous or acrosomales enzymes were correlated with oocyte cytoskeleton disruption through an aberrant accumulation of microtubules in the cortex of the oocyte.

   In addition to the morphological and ultrastructural alterations in the oocyte, the incorporation of the acrosome may result in a lack of nuclear activation of the oocyte. Kasai et al. reported that the completion of oocyte meiosis occur faster if the sperm was released from the acrosome. Similarly, an increase in fertilization rate after ICSI with acrosome reacted sperm was observed in pigs. The study by Morozumi et al. also demonstrated that the induction of the acrosome reaction of sperm from several species prior to ICSI resulted in an acceleration of oocyte activation, which was manifest in human spermatozoa. This was evidenced by the significant differences between the profiles of calcium oscillations after ICSI with acrosome-intact or acrosome-reacted sperm. Calcium waves recorded in oocytes injected with acrosome-reacted spermatozoa were characterized by an early onset and amplitude and a higher frequency. In contrast, the calcium response was abnormally delayed in oocytes injected with acrosome-intact sperm.

   Thus, altered calcium oscillations, the "key" oocyte activation signals during ICSI, is the cause of abnormal pre-implantation embryo development to the blastocyst stage. Indeed, the proportion of live healthy mice births is increased from 40% to 71%, when intact or acrosome-reacted sperm are microinjected, respectively .

   These same studies have also shown two things:
   * The introduction of acrosomal material is more harmful when the quantity is large compared to the oocyte volume. There is therefore interest in systematically reducing the amount of material introduced into the oocyte cytoplasm to improve embryonic development.
   * The second thing is that the induction of the acrosome reaction before ICSI greatly improves embryonic development and therefore the number of babies born from embryo transfer.

   Although ICSI in human gives very satisfactory results, the rate of infants obtained by embryo is lower than after IVF embryos transfer. Hence, there is a possibility of improving the results of ICSI by induction of the acrosome reaction prior to microinjection.

   After several studies we used incubation of spermatozoa with the follicular fluid (FF) of the partner to induce the spermatozoa acrosome reaction (Karim Rahal, 2011 Master Thesis 2). FF is indeed a potent inducer of the AR. There is no problem of traceability since the FF of the patient is used only for the sperm of her husband. This technic can be applied to the poorest semen. Finally, the technique is used in a very easy routine, since the follicular fluid is always recovered during oocyte retrieval and thus available.
2. Hypothesis A preliminary study was run in human on microinjection of spermatozoa that were selected for their acrosomal status by birefringence microscopy. It showed that it improves the implantation rate from 24,4 % to 39 % . We therefore hypothesize that the improvement in the implantation rate of embryos obtained by ICSI after acrosomal induction as well as the reduction of miscarriage rate may result in improved clinical pregnancy outcome and birth rates of about 10 %.

ELIGIBILITY:
Inclusion Criteria:

* Couples involved in an ICSI program
* First attempt only
* Cohort with at least 6 oocytes

Exclusion Criteria:

* No social security number
* No signed consent form
* Surgically retrieved sperm

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 620 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
number of early pregnancy termination | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Background] Lacham-Kaplan O, Trounson A. Intracytoplasmic sperm injection in mice: increased fertilization and development to term after induction of the acrosome reaction. Hum Reprod. 1995 Oct;10(10):2642-9. doi: 10.1093/oxfordjournals.humrep.a135760. PMID 8567785
- [Background] Roldan ER. Better intracytoplasmic sperm injection without sperm membranes and acrosome. Proc Natl Acad Sci U S A. 2006 Nov 21;103(47):17585-6. doi: 10.1073/pnas.0608752103. Epub 2006 Nov 13. No abstract available. PMID 17101960
- [Background] Morozumi K, Shikano T, Miyazaki S, Yanagimachi R. Simultaneous removal of sperm plasma membrane and acrosome before intracytoplasmic sperm injection improves oocyte activation/embryonic development. Proc Natl Acad Sci U S A. 2006 Nov 21;103(47):17661-6. doi: 10.1073/pnas.0608183103. Epub 2006 Nov 7. PMID 17090673